CLINICAL TRIAL: NCT03393585
Title: Respiratory Rates - Accuracy of Contact-free Monitoring of Respiratory Rates in the Triage Setting of an Emergency Department
Brief Title: Respiratory Rates - Accuracy of Contact-free Monitoring of Respiratory Rates
Status: Completed | Type: Observational
Sponsor: Christian Nickel (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Christian Nickel, PD MD, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: Resprate 2017; EKNZ 2017-01583 (Other: swissethics)
Record Dates: First submitted 2017-12-21; First posted 2018-01-08 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Emergencies; Tachypnea
Keywords: Respiratory Rates
MeSH Terms: conditions — Emergencies; Tachypnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: touchless vital signs monitoring — We measure Respiratory Rates in the Triage of Patients entering an Emergency Department by three different methods.

SUMMARY:
Respiratory rate is an important predictor for many clinical outcomes in Emergency Medicine. Nevertheless it's measurement is often omitted as it is time-consuming and cumbersome. It is the only vital sign that is not routinely assessed by a device. In a pilot study was showed that a camera based monitoring system measures reliably respiratory rates in healthy volunteers.

The goal of this study is to test the accuracy of the same system in real patients in the triage setting of an Emergency Department (ED).

DETAILED DESCRIPTION:
For triage of emergency patients at the Emergency Department of the University Hospital Basel the emergency severity index (ESI) is used. At decision point "D" in the ESI-algorithm vital signs such as respiratory rate, heart rate and oxygen saturation are needed.

According to the guidelines the respiratory rate is visually counted for one minute (WHOrecommendation) by a triage nurse.

Simultaneously in addition to the visual counting, it is planned to measure the same vital sign as part of our study also through a camera-based prototype application (CBPA) and capnography as a gold standard.

Hence the triage process is not prolongated through our study, only completed and a guideline compliant procedure is ensured which is only performed in a relatively low percentage in the ED of the University Hospital Basel. Clinical decisions are exclusively based on the actual clinical standard of visual counting and are not influenced by the measurements of our study.

For the capnography, which were considered as the most accurate method, the patient wears a nasal sample line (Philips® Heartstart MRx mit Philips® Smart CapnoLine™PlusO2Long Oral/Nasal Sample Line).

The CBPA system consists of a notebook (HP Zbook 15 G3, S/N: CND705IXT6), USB-camera with lens (Tamron CCTV lens, CE 4402789484; UI3060 camera, 20170329-E347840), USB-harddrive (Western digital R/N D8B, S/N: WXA1E661J0XJ) to save the signals and an implement camera-based algorithm for extraction of breathing signals. The camera is pointing towards the torso of the patient to display it on the screen in a real-time application. The software is able to detect the respiratory-specific chest movements and generates a respiratory wave on the computer. From the configuration and frequency of these respiratory waves the software calculates the respiratory rate. No videos are recorded.

The data is acquired in a standardised protocol and stored coded in an Access®-database. To prevent potential bias the vital signs will be written down in the following order: 1. RR by visual counting 2. RR by CBPA 3. RR by capnography. The measurements take place in rooms of the ED which are designated to triage emergency patients.

As possible confounders sex, age and BMI are registered.

ELIGIBILITY:
Inclusion Criteria:

* All walk-in patients older than 18 with a presumed ESI score of 2-3 presenting to the ED of the University Hospital of Basel will be eligible for inclusion.

Exclusion Criteria:

* Excluded will be (1) patients brought in by ambulance or helicopter, (2) unstable patients needing immediate medical treatment, (3) confused, restless, deaf patients having difficulty to follow the study instructions (4) Clear signs of refusal to participate the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will contain patients running through triage of the Emergency Department with an indication for vital sign assessment. The data will only be collected in the University Hospital of Basel.
Sampling Method: Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2017-12-23 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Specificity and sensitivity of the camera based prototype application (CBPA) | 1 year
  In this study respiratory rates are obtained by 3 methods. 1. Camera based measurement, 2. with capnography and 3. with the WHO criterion standard of counting breaths for 1 Minute (18 measurements in whole). We want to study the Specificity and sensitivity of the CBPA compared to the gold standard (capnography)

SECONDARY OUTCOMES:
Upgrade of patient's ESI level due to CBPA (from Level 3 to 2) | 1 year
  Number of Patients with a RR measured by CBPA higher than 20 leading to an upgrade at decision Point D of the Triage algorithm (ESI)

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Nickel, PD Dr. med, Principal Investigator — Emergency Department, University Hospital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodgetts TJ, Kenward G, Vlachonikolis IG, Payne S, Castle N. The identification of risk factors for cardiac arrest and formulation of activation criteria to alert a medical emergency team. Resuscitation. 2002 Aug;54(2):125-31. doi: 10.1016/s0300-9572(02)00100-4. PMID 12161291
- [Background] Strauss R, Ewig S, Richter K, Konig T, Heller G, Bauer TT. The prognostic significance of respiratory rate in patients with pneumonia: a retrospective analysis of data from 705,928 hospitalized patients in Germany from 2010-2012. Dtsch Arztebl Int. 2014 Jul 21;111(29-30):503-8, i-v. doi: 10.3238/arztebl.2014.0503. PMID 25142073
- [Background] Bone RC, Sprung CL, Sibbald WJ. Definitions for sepsis and organ failure. Crit Care Med. 1992 Jun;20(6):724-6. doi: 10.1097/00003246-199206000-00002. No abstract available. PMID 1597021
- [Background] Brabrand M, Havshoj U, Graham CA. Validation of the qSOFA score for identification of septic patients: A retrospective study. Eur J Intern Med. 2016 Dec;36:e35-e36. doi: 10.1016/j.ejim.2016.09.004. Epub 2016 Sep 15. No abstract available. PMID 27640097
- [Background] Mower WR, Sachs C, Nicklin EL, Safa P, Baraff LJ. A comparison of pulse oximetry and respiratory rate in patient screening. Respir Med. 1996 Nov;90(10):593-9. doi: 10.1016/s0954-6111(96)90017-7. PMID 8959116
- [Background] Subbe CP, Kruger M, Rutherford P, Gemmel L. Validation of a modified Early Warning Score in medical admissions. QJM. 2001 Oct;94(10):521-6. doi: 10.1093/qjmed/94.10.521. PMID 11588210
- [Background] Goldhill DR, White SA, Sumner A. Physiological values and procedures in the 24 h before ICU admission from the ward. Anaesthesia. 1999 Jun;54(6):529-34. doi: 10.1046/j.1365-2044.1999.00837.x. PMID 10403864
- [Background] Grossmann FF, Nickel CH, Christ M, Schneider K, Spirig R, Bingisser R. Transporting clinical tools to new settings: cultural adaptation and validation of the Emergency Severity Index in German. Ann Emerg Med. 2011 Mar;57(3):257-64. doi: 10.1016/j.annemergmed.2010.07.021. Epub 2010 Oct 16. PMID 20952097
- [Background] Hossein Nejad H, Banaie M, Seyedhosseini Davarani SH, Khazaeipour Z. Evaluation of the Significance of Vital Signs in the Up-Triage of Patients Visiting Emergency Department from Emergency Severity Index Level 3 to 2. Acta Med Iran. 2016 Jun;54(6):366-9. PMID 27306342
- [Background] Hogan J. Why don't nurses monitor the respiratory rates of patients? Br J Nurs. 2006 May 11-24;15(9):489-92. doi: 10.12968/bjon.2006.15.9.21087. PMID 16723921
- [Background] Lovett PB, Buchwald JM, Sturmann K, Bijur P. The vexatious vital: neither clinical measurements by nurses nor an electronic monitor provides accurate measurements of respiratory rate in triage. Ann Emerg Med. 2005 Jan;45(1):68-76. doi: 10.1016/j.annemergmed.2004.06.016. PMID 15635313
- [Background] Edmonds ZV, Mower WR, Lovato LM, Lomeli R. The reliability of vital sign measurements. Ann Emerg Med. 2002 Mar;39(3):233-7. doi: 10.1067/mem.2002.122017. PMID 11867974
- [Background] Folke M, Cernerud L, Ekstrom M, Hok B. Critical review of non-invasive respiratory monitoring in medical care. Med Biol Eng Comput. 2003 Jul;41(4):377-83. doi: 10.1007/BF02348078. PMID 12892358
- [Background] Becker C, Achermann S, Rocque M, Kirenko I, Schlack A, Dreher-Hummel T, Zumbrunn T, Bingisser R, Nickel CH. Camera-based measurement of respiratory rates is reliable. Eur J Emerg Med. 2018 Dec;25(6):416-422. doi: 10.1097/MEJ.0000000000000476. PMID 28574856
- [Background] Flahault A, Cadilhac M, Thomas G. Sample size calculation should be performed for design accuracy in diagnostic test studies. J Clin Epidemiol. 2005 Aug;58(8):859-62. doi: 10.1016/j.jclinepi.2004.12.009. PMID 16018921
- [Derived] Caspar M, Dutilh G, Achermann S, Bingisser R, Nickel CH. Contact-Free Monitoring of Pulse Rate For Triage of Patients Presenting to the Emergency Department. J Emerg Med. 2021 Dec;61(6):649-657. doi: 10.1016/j.jemermed.2021.07.005. Epub 2021 Aug 30. PMID 34474932
- [Derived] Achermann S, Caspar M, Wirth C, Becker C, Rocque M, Kirenko I, Schlack A, Dutilh G, Bingisser R, Nickel CH. Contact-free monitoring of respiratory rates for triage of patients presenting to the emergency department. Resuscitation. 2019 Apr;137:154-155. doi: 10.1016/j.resuscitation.2019.01.041. Epub 2019 Feb 18. No abstract available. PMID 30790695